CLINICAL TRIAL: NCT02452307
Title: Prospective Randomized Trial of Peptide-specific Vaccination in HLA-A*02 Positive Prostate Carcinoma Patients With Biochemical Recurrence After Radical Prostatectomy
Brief Title: Peptide-specific Vaccination in HLA-A*02 Positive Patients With Biochemical Recurrence After Radical Prostatectomy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 167/2003
Record Dates: First submitted 2015-04-14; First posted 2015-05-22 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Recurrent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Protein Subunit Vaccines; montanide ISA 51; Granulocyte-Macrophage Colony-Stimulating Factor; Imiquimod; RNA, Messenger; somatostatin, protamine zinc-; Hyperthermia, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Peptide vaccine (Experimental): Subcutaneous application of Prostate-specific peptide vaccine compound emulsified in Montanide ISA-51
  Interventions: Biological: Peptide vaccine; Drug: Montanide ISA-51
- Peptide vaccine + GM-CSF (Experimental): Subcutaneous application of Prostate-specific peptide vaccine compound emulsified in Montanide ISA-51 in combination with Granulocyte macrophage colony stimulating factor (GM-CSF)
  Interventions: Biological: Peptide vaccine; Drug: Montanide ISA-51; Drug: Granulocyte macrophage colony stimulating factor (GM-CSF)
- Peptide vaccine + local hyperthermia (Experimental): Subcutaneous application of Prostate-specific peptide vaccine compound emulsified in Montanide ISA-51 in combination with local hyperthermia
  Interventions: Biological: Peptide vaccine; Drug: Montanide ISA-51; Procedure: local hyperthermia
- Peptide vaccine + Imiquimod (Experimental): Subcutaneous application of Prostate-specific peptide vaccine compound emulsified in Montanide ISA-51 in combination with Imiquimod
  Interventions: Biological: Peptide vaccine; Drug: Montanide ISA-51; Drug: Imiquimod
- Peptide vaccine + mRNA/Protamin (Experimental): Subcutaneous application of Prostate-specific peptide vaccine compound emulsified in Montanide ISA-51 in combination with mRNA/Protamin
  Interventions: Biological: Peptide vaccine; Drug: Montanide ISA-51; Drug: mRNA; Drug: Protamin

INTERVENTIONS:
Biological: Peptide vaccine — subcutaneous
Drug: Montanide ISA-51 — subcutaneous
Drug: Granulocyte macrophage colony stimulating factor (GM-CSF) — intradermal
  Arms: Peptide vaccine + GM-CSF
Drug: Imiquimod — epicutaneous
  Arms: Peptide vaccine + Imiquimod
Drug: mRNA — subcutaneous
  Arms: Peptide vaccine + mRNA/Protamin
Drug: Protamin — subcutaneous
  Arms: Peptide vaccine + mRNA/Protamin
Procedure: local hyperthermia
  Arms: Peptide vaccine + local hyperthermia

SUMMARY:
The study evaluates the prostate-specific antigen (PSA) response in HLA-A*02 positive patients with biochemical recurrence after radical prostatectomy treated with a prostate-specific peptide vaccine in combination with different immune-adjuvants.

DETAILED DESCRIPTION:
Patients with a biochemical recurrence after initial therapy can be included.

ELIGIBILITY:
Inclusion Criteria:

* biochemical recurrence after Radical Prostatectomy
* no clinical metastases in CT or bone scan
* HLA-Type: HLA-A*02 positive
* Karnofsky-Performance-Index >70
* Age >45 / <80 years
* no prior or ongoing hormonal therapy
* no ongoing radiation therapy
* Serum-Creatinine <2mg/dl; Bilirubin: <2gm/dl
* no history of allergy or chronic obstructive lung disease (COLD)

Exclusion Criteria:

* Patients unable to consent
* Karnofsky-Performance-Index <70
* known allergy or COLD
* presence of secondary malignancy
* prior or ongoing hormonal treatment
* ongoing radiotherapy
* immunosuppressive medication
* seizure

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-04; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Immune Response at day 70 | Days 0-70
  Immune Response, as measured by the change of in vitro and in vivo T cell response from baseline at day 0 to day 70

SECONDARY OUTCOMES:
Tolerability | Days 0-420
  Tolerability, as measured by number of Participants with Adverse Events
Treatment response | Months 0-60
  Treatment response, from date of randomization until the date of first documented progression as measured by PSA-value

CONTACTS AND LOCATIONS:
Overall Officials: Arnulf Stenzl, Prof., Principal Investigator — Department of Urology, University of Tuebingen